CLINICAL TRIAL: NCT02098252
Title: Treatment of Brain AVMs (TOBAS) Study: A Randomized Controlled Trial and Registry
Brief Title: Treatment of Brain AVMs (TOBAS) Study
Acronym: TOBAS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Centre Hospitalier Régional et Universitaire de Brest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13.315
Record Dates: First submitted 2014-03-25; First posted 2014-03-27 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Unruptured Brain Arteriovenous Malformation; Ruptured Brain Arteriovenous Malformation; Arteriovenous Malformations; AVM; BAVM
Keywords: brain arteriovenous malformation; Arteriovenous Malformations; AVM; BAVM; Stroke; Intracranial Hemorrhage; Congenital Abnormalities; Aneurysm; Vascular Malformations; Cardiovascular Abnormalities; Cardiovascular Diseases; Vascular Diseases
MeSH Terms: conditions — Arteriovenous Malformations; Stroke; Intracranial Hemorrhages; Congenital Abnormalities; Aneurysm; Vascular Malformations; Cardiovascular Abnormalities; Cardiovascular Diseases; Vascular Diseases | interventions — Neurosurgical Procedures; Radiotherapy; Embolization, Therapeutic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Interventional therapy (Active Comparator): Interventional therapies include:
  neurosurgery (surgical resection when the lesion is considered by a multidisciplinary team to be safely 'operable'); radiation therapy (when the AVM is smaller than 3 cm, and considered to not be safely 'operable'); radiosurgery, alone or in combination, with or without endovascular procedure; curative embolization (when the lesion is considered curable by embolization).
  Patients with AVMs that the multidisciplinary team judges could potentially benefit from endovascular treatment prior to surgical resection or radiation therapy will then also be pre-randomly allocated to embolization or to no embolization.
  Interventions: Procedure: Neurosurgery; Radiation: Radiation therapy; Procedure: Embolization
- Conservative management (medical management) (No Intervention): The conservative, or medical management arm, involves pharmacological therapy as deemed appropriate for medical symptoms as determined by the treating investigator. Should patients in the conservative management arm develop hemorrhage or infarction related to their AVM, they then potentially become candidates for interventional therapy.

INTERVENTIONS:
Procedure: Neurosurgery — Surgical resection to be used when the lesion is considered by a multidisciplinary team to be safely 'operable'.
  Arms: Interventional therapy
Radiation: Radiation therapy — when the AVM is smaller than 3 cm, and considered to not be safely 'operable'.
  Arms: Interventional therapy
Procedure: Embolization — Curative embolization, when the lesion is considered curable by embolization.
  Arms: Interventional therapy

SUMMARY:
The objectives of this study and registry are to offer the best management possible for patients with brain arteriovenous malformations (AVMs) (ruptured or unruptured) in terms of long-term outcomes, despite the presence of uncertainty. Management may include interventional therapy (with endovascular procedures, neurosurgery, or radiotherapy, alone or in combination) or conservative management.

The trial has been designed to test a) whether medical management or interventional therapy will reduce the risk of death or debilitating stroke (due to hemorrhage or infarction) by an absolute magnitude of about 15% (over 10 years) for unruptured AVMs (from 30% to 15%); and, b) to test if endovascular treatment can improve the safety and efficacy of surgery or radiation therapy by at least 10% (80% to 90%).

As for the nested trial on the role of embolization in the treatment of Brain AVMs by other means: the pre-surgical or pre-radiosurgery embolization of cerebral AVMs can decrease the number of treatment failures from 20% to 10%. In addition,embolization of cerebral AVMs can be accomplished with an acceptable risk, defined as permanent disabling neurological complications of 8%.

DETAILED DESCRIPTION:
Intracranial arteriovenous malformations (AVMs) are relatively uncommon but increasingly discovered lesions that can lead to significant neurological disability or death.1 Population-based data suggest that the annual incidence of discovery of a symptomatic AVM is approximately 1.1 per 100 000 population.7. AVMs commonly present following an intracranial hemorrhage or seizure, although with contemporary brain imaging techniques, an increasing number of incidental lesions are found.2

Intracranial AVMs are typically diagnosed before the age of 40 years old, with more than 50% of patients presenting following an intracranial hemorrhage, the most feared sequelae of harbouring an AVM.3 An AVM-related seizure is reported as the presenting feature in 20-25% of cases4, 5 and although these can sometimes be successfully managed with anti-epileptic agents, some AVMs lead to intractable seizures in spite of medication. Other presentations include headaches, focal neurological deficits, or pulsatile tinnitus.1

The available natural history studies indicate an overall risk of initial hemorrhage of approximately 2% to 4% per year, although the long-term consequences in terms of the probability of death or long-term disability following intracranial hemorrhage remains unclear.6-8 Mortality from the first hemorrhage has been reported to occur between 10-30% of patients with a ruptured AVM, although some more recent data suggest that the mortality rate may be lower and only 10-20% of survivors have long-term disability.9-11 Hemorrhagic presentation is considered the most reliable risk factor for a repeat hemorrhage.6, 8 Unfortunately, the natural history data available is not of sufficient quality (Level V) to support making management recommendations.

Over the last decade, there have been substantial developments in the management of intracranial AVMs. There has been an evolution of microsurgical as well as endovascular and radiosurgical techniques to treat these lesions. As the management options have evolved, individual and combined modality treatment protocols have been developed in different institutions for the management of AVMs. Current interventional therapy for brain arteriovenous malformations (BAVMs) is varied and includes open neurosurgical resection, radiosurgery, and endovascular management, either alone or in combination. The choice of management is largely dependent on the decisions of the local physicians that make up the treatment team, and a recent survey has demonstrated substantial variability in decision-making for almost all AVMs.12

Interventional therapies, when they are performed, are assumed to decrease the risk of initial or subsequent hemorrhage and therefore lead to better long-term outcomes, an assumption that has yet to be proven.

Although the question of which AVM treatment modality is the most appropriate first choice (surgery, radiosurgery, or embolization) remains controversial, consensus can be reached in several circumstances. Surgical evacuation of a hematoma exerting significant mass effect is an uncontested appropriate management, although many patients with a hemorrhagic presentation do not necessarily meet this threshold for surgical indication. Almost all other management choices remain debatable.13, 14 A systematic review has proposed that approximately 7.1% of surgical candidates, 6.6% of endovascular candidates, and 5.1% of radiosurgical candidates were facing permanent neurological deficits after treatment.15 The epidemiological study of Davies et al, using the Nationwide Inpatient Sample (NIS) data base and surrogates such as location at discharge, showed worse outcomes for surgical and endovascular management of both ruptured and unruptured AVMs.16

Current choices of interventional therapy for brain arteriovenous malformations are varied, with decisions made on a case-by-case basis, by the local clinical team. Often these decisions will change as the results of one particular attempted treatment modality become available. All interventional therapies are performed with the assumption that they will decrease the risk of initial or subsequent hemorrhage and lead to better long-term patient outcomes. Despite these laudable goals, there is no reliable evidence that interventional management of unruptured bAVMs is beneficial, and in patients judged to need interventional therapy, such as those patients presenting with ruptures, there is no randomized evidence that embolization is beneficial. Although no clinical trial data exist on the effect of interventional therapy even after AVM hemorrhage, the most contentious issue at present is whether interventional therapy should be considered for patients with incidentally discovered AVMs, whose lesions have not bled. In patients with unruptured AVMs, the best management strategy remains unknown, and interventions should be proposed only in the context of a randomized trial.

The potential role of embolization: Although endovascular AVM embolization can occasionally eradicate lesions without surgery or radiation therapy in selected cases, and although embolization may potentially improve the safety and efficacy of surgical or radiosurgical treatments in some other cases, it remains a contentious issue whether it is worth accepting the additional risks of endovascular treatment for a greater overall benefit for patients with brain AVMs that are treatable by surgery or radiation therapy. Some series have reported satisfactory results.20 It is possible that the overall morbidity and mortality of the combined interventional management strategy is increased when embolization is added to a surgical or radiosurgical procedure.17 Therefore, pre-surgical or pre-radiosurgical embolization can be offered, but only as a randomized allocation between embolization and no embolization, within the context of a trial.

Primary objective: In the spirit of care trials, the primary objective of the trial and accompanying registry is to offer the best management possible for patients with brain AVMs (ruptured or unruptured) in terms of long-term outcomes, despite the presence of uncertainty. Management may include interventional therapy (neurosurgery, or radiosurgery, alone or in combination, with or without endovascular procedures, alone or combined) or conservative management. An expert multidisciplinary study group will review patients on an individual basis to determine eligibility for the trial or registry parts of the study. The trial has been designed to test whether conservative management or interventional therapy will reduce the risk of disabling stroke or death.

Secondary objectives: To determine if interventional management is effective in the prevention of neurological events during 10 years. To determine the morbidity and mortality related to therapy. To follow-up and record the neurological events and the neurological status of all patients with brain AVMs recruited and managed in our institutions, regardless of management strategy chosen.

Hypotheses

A) Randomized comparison of interventional treatment and conservative management:

Primary hypothesis: Treatment of cerebral AVMs can decrease the number of disabling neurological events caused by the presence of the AVM (excluding peri-operative complications) from 30 to 15% within 10 years. (n = 266 minima) Secondary hypothesis: Treatment of cerebral AVMs can be accomplished with an acceptable up-front risk, defined as the occurrence of a permanent disabling neurological complication in less than 15% of patients)

B) Nested trial on the Role of embolization in the treatment of Brain AVMs by other means Primary hypothesis: Pre-surgical or pre-radiosurgery embolization of cerebral AVMs can decrease the number of treatment failures (failure to achieve angiographic cure) from 20% to 10% (n= 440).

Secondary hypothesis: Embolization of cerebral AVMs can be accomplished with an acceptable risk, defined as permanent disabling neurological complications of 8% (3.4 to 12.6%, 95% C.I.).

The study design is a prospective, multi-center, randomized, controlled trial and registry. Treatment assignment will not be masked; Interim study results will be kept confidential. The primary outcome is the composite event of death from any cause or disabling stroke (hemorrhage or infarction revealed by imaging and resulting in mRS >2). Functional outcome status will be measured by the Rankin Scale, a widely used outcome measure for stroke. The secondary measures of outcome include adverse events, ruptures, and angiographic occlusion of the lesion.

ELIGIBILITY:
Inclusion Criteria:

* Any patient with a brain AVM

Exclusion Criteria:

* Hemorrhagic presentation with mass effect requiring surgical management. In these cases, if a residual AVM is found after the initial surgery, the patient could then be a candidate for TOBAS.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2014-05; Primary Completion 2035-01 (Estimated); Study Completion 2036-01 (Estimated)

PRIMARY OUTCOMES:
composite event of death from any cause or disabling stroke | up to 10 years post-treatment (or randomization)
  death or disabling stroke due to hemorrhage or infarction as revealed by imaging and resulting in mRS >2.

SECONDARY OUTCOMES:
occurrence of any neurological event | within 10 years following treatment (or after randomization)
Permanent disabling peri-operative complications | within 31 days post-treatment
  The incidence of permanent (more than 3 months) disabling (mRS >2) peri-operative (within 31 days) complications

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Roy, MD, Principal Investigator — CHUM-Montreal
Locations (30):
- United States (3):
  - Mayo Clinic in Jacksonville FL, Jacksonville, Florida
  - Boston Medical Center, Boston, Massachusetts
  - University of New Mexico Health Sciences Center, Albuquerque, New Mexico
- Brazil (2):
  - Hospital Geral de Fortaleza, Fortaleza
  - Universidade Federal de Sǎo Paulo, São Paulo
- Canada (2):
  - University of Alberta Hospital, Edmonton, Alberta
  - Klink, Ruby, Montreal, Quebec
- Instituto de Neurocirugia Dr. A. Asenjo, Santiago, Chile
- Universidad Autonoma de Bucaramanga, Bucaramanga, Colombia
- France (21):
  - CHRU de Brest (Brest University Hospital), Brest, Brittany Region
  - Centre Hospit Régional Universitaire de Besançon, Besançon
  - Centre Hospitalier Universitaire de Bordeaux, Bordeaux
  - Centre Hospitalier Universitaire de Caen, Caen
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - CHU Dijon Bourgogne, Dijon
  - Hôpital Bicêtre AP-HP, Le Kremlin-Bicêtre
  - CHU Limoges, Limoges
  - Centre Hospitalier Universitaire de Lyon, Lyon
  - Assistance Publique - Hôpitaux de Marseille, Marseille
  - Centre Hospitalier Universitaire de Montpellier, Montpellier
  - Centre Hospitalier Régional Universitaire de Nancy, Nancy
  - Centre Hospitalier Universitaire de Nantes, Nantes
  - Hôpital Universitaire Pitié-Salpêtrière, Paris
  - Fondation Ophtalmologique Rothschild, Paris
  - Centre Hospitalier Sainte-Anne, Paris
  - Centre Hospitalier Universitaire de Rennes, Rennes
  - Centre Hospitalier Universitaire Hôpitaux de Rouen, Rouen
  - Les Hôpitaux Universitaires de Strasbourg, Strasbourg
  - Centre Hospitalier Universitaire de Toulouse, Toulouse
  - Centre Hospitalier Régional Universitaire de Tours, Tours

REFERENCES:
- [Background] Fleetwood IG, Steinberg GK. Arteriovenous malformations. Lancet. 2002 Mar 9;359(9309):863-73. doi: 10.1016/S0140-6736(02)07946-1. PMID 11897302
- [Background] Wedderburn CJ, van Beijnum J, Bhattacharya JJ, Counsell CE, Papanastassiou V, Ritchie V, Roberts RC, Sellar RJ, Warlow CP, Al-Shahi Salman R; SIVMS Collaborators. Outcome after interventional or conservative management of unruptured brain arteriovenous malformations: a prospective, population-based cohort study. Lancet Neurol. 2008 Mar;7(3):223-30. doi: 10.1016/S1474-4422(08)70026-7. Epub 2008 Feb 1. PMID 18243054
- [Background] Brown RD Jr, Wiebers DO, Torner JC, O'Fallon WM. Frequency of intracranial hemorrhage as a presenting symptom and subtype analysis: a population-based study of intracranial vascular malformations in Olmsted Country, Minnesota. J Neurosurg. 1996 Jul;85(1):29-32. doi: 10.3171/jns.1996.85.1.0029. PMID 8683279
- [Background] Brown RD Jr, Wiebers DO, Forbes G, O'Fallon WM, Piepgras DG, Marsh WR, Maciunas RJ. The natural history of unruptured intracranial arteriovenous malformations. J Neurosurg. 1988 Mar;68(3):352-7. doi: 10.3171/jns.1988.68.3.0352. PMID 3343606
- [Background] Wilkins RH. Natural history of intracranial vascular malformations: a review. Neurosurgery. 1985 Mar;16(3):421-30. doi: 10.1227/00006123-198503000-00026. PMID 3885072
- [Background] da Costa L, Wallace MC, Ter Brugge KG, O'Kelly C, Willinsky RA, Tymianski M. The natural history and predictive features of hemorrhage from brain arteriovenous malformations. Stroke. 2009 Jan;40(1):100-5. doi: 10.1161/STROKEAHA.108.524678. Epub 2008 Nov 13. PMID 19008469
- [Background] Gross BA, Du R. Natural history of cerebral arteriovenous malformations: a meta-analysis. J Neurosurg. 2013 Feb;118(2):437-43. doi: 10.3171/2012.10.JNS121280. Epub 2012 Nov 30. PMID 23198804
- [Background] Hernesniemi JA, Dashti R, Juvela S, Vaart K, Niemela M, Laakso A. Natural history of brain arteriovenous malformations: a long-term follow-up study of risk of hemorrhage in 238 patients. Neurosurgery. 2008 Nov;63(5):823-9; discussion 829-31. doi: 10.1227/01.NEU.0000330401.82582.5E. PMID 19005371
- [Background] Hartmann A, Mast H, Mohr JP, Koennecke HC, Osipov A, Pile-Spellman J, Duong DH, Young WL. Morbidity of intracranial hemorrhage in patients with cerebral arteriovenous malformation. Stroke. 1998 May;29(5):931-4. doi: 10.1161/01.str.29.5.931. PMID 9596237
- [Background] Hartmann A, Mast H, Mohr JP, Pile-Spellman J, Connolly ES, Sciacca RR, Khaw A, Stapf C. Determinants of staged endovascular and surgical treatment outcome of brain arteriovenous malformations. Stroke. 2005 Nov;36(11):2431-5. doi: 10.1161/01.STR.0000185723.98111.75. Epub 2005 Oct 13. PMID 16224095
- [Background] Hartmann A, Stapf C, Hofmeister C, Mohr JP, Sciacca RR, Stein BM, Faulstich A, Mast H. Determinants of neurological outcome after surgery for brain arteriovenous malformation. Stroke. 2000 Oct;31(10):2361-4. doi: 10.1161/01.str.31.10.2361. PMID 11022064
- [Background] Cockroft KM, Chang KE, Lehman EB, Harbaugh RE. AVM Management Equipoise Survey: physician opinions regarding the management of brain arteriovenous malformations. J Neurointerv Surg. 2014 Dec;6(10):748-53. doi: 10.1136/neurintsurg-2013-011030. Epub 2013 Dec 6. PMID 24319022
- [Background] Cockroft KM. Unruptured brain arteriovenous malformations should be treated conservatively: no. Stroke. 2007 Dec;38(12):3310-1. doi: 10.1161/STROKEAHA.107.504613. Epub 2007 Oct 25. No abstract available. PMID 17962584
- [Background] Stapf C, Mohr JP. Unruptured brain arteriovenous malformations should be treated conservatively: yes. Stroke. 2007 Dec;38(12):3308-9. doi: 10.1161/STROKEAHA.107.504605. Epub 2007 Oct 25. No abstract available. PMID 17962585
- [Background] van Beijnum J, van der Worp HB, Buis DR, Al-Shahi Salman R, Kappelle LJ, Rinkel GJ, van der Sprenkel JW, Vandertop WP, Algra A, Klijn CJ. Treatment of brain arteriovenous malformations: a systematic review and meta-analysis. JAMA. 2011 Nov 9;306(18):2011-9. doi: 10.1001/jama.2011.1632. PMID 22068993
- [Background] Davies JM, Yanamadala V, Lawton MT. Comparative effectiveness of treatments for cerebral arteriovenous malformations: trends in nationwide outcomes from 2000 to 2009. Neurosurg Focus. 2012 Jul;33(1):E11. doi: 10.3171/2012.5.FOCUS12107. PMID 22746228
- [Background] Morgan MK, Davidson AS, Koustais S, Simons M, Ritson EA. The failure of preoperative ethylene-vinyl alcohol copolymer embolization to improve outcomes in arteriovenous malformation management: case series. J Neurosurg. 2013 May;118(5):969-77. doi: 10.3171/2012.11.JNS112064. Epub 2013 Jan 25. PMID 23350776
- [Background] Pierot L, Fiehler J, Cognard C, Soderman M, Spelle L. Will a randomized trial of unruptured brain arteriovenous malformations change our clinical practice? AJNR Am J Neuroradiol. 2014 Mar;35(3):416-7. doi: 10.3174/ajnr.A3867. Epub 2014 Jan 16. No abstract available. PMID 24436345
- [Background] Raymond J; TEAM collaborative group. Reflections on the TEAM trial: why clinical care and research should be reconciled. Can J Neurol Sci. 2011 Mar;38(2):198-202. doi: 10.1017/s0317167100011343. PMID 21320821
- [Background] Saatci I, Geyik S, Yavuz K, Cekirge HS. Endovascular treatment of brain arteriovenous malformations with prolonged intranidal Onyx injection technique: long-term results in 350 consecutive patients with completed endovascular treatment course. J Neurosurg. 2011 Jul;115(1):78-88. doi: 10.3171/2011.2.JNS09830. Epub 2011 Apr 8. PMID 21476804
- [Background] Spetzler RF, Martin NA. A proposed grading system for arteriovenous malformations. J Neurosurg. 1986 Oct;65(4):476-83. doi: 10.3171/jns.1986.65.4.0476. PMID 3760956
- [Derived] Raymond J, Gentric JC, Magro E, Nico L, Bacchus E, Klink R, Cognard C, Januel AC, Sabatier JF, Iancu D, Weill A, Roy D, Bojanowski MW, Chaalala C, Barreau X, Jecko V, Papagiannaki C, Derrey S, Shotar E, Cornu P, Eker OF, Pelissou-Guyotat I, Piotin M, Aldea S, Beaujeux R, Proust F, Anxionnat R, Costalat V, Corre ML, Gauvrit JY, Morandi X, Brunel H, Roche PH, Graillon T, Chabert E, Herbreteau D, Desal H, Trystram D, Barbier C, Gaberel T, Nguyen TN, Viard G, Gevry G, Darsaut TE; TOBAS Collaborative Group; Collaborators in the TOBAS Collaborative Group. Endovascular treatment of brain arteriovenous malformations: clinical outcomes of patients included in the registry of a pragmatic randomized trial. J Neurosurg. 2022 Oct 28;138(5):1393-1402. doi: 10.3171/2022.9.JNS22987. Print 2023 May 1. PMID 37132535
- [Derived] Darsaut TE, Magro E, Bojanowski MW, Chaalala C, Nico L, Bacchus E, Klink R, Iancu D, Weill A, Roy D, Sabatier JF, Cognard C, Januel AC, Pelissou-Guyotat I, Eker O, Roche PH, Graillon T, Brunel H, Proust F, Beaujeux R, Aldea S, Piotin M, Cornu P, Shotar E, Gaberel T, Barbier C, Corre ML, Costalat V, Jecko V, Barreau X, Morandi X, Gauvrit JY, Derrey S, Papagiannaki C, Nguyen TN, Abdalkader M, Tawk RG, Huynh T, Viard G, Gevry G, Gentric JC, Raymond J; TOBAS Collaborative Group; List of participating TOBAS centers and physicians. Surgical treatment of brain arteriovenous malformations: clinical outcomes of patients included in the registry of a pragmatic randomized trial. J Neurosurg. 2022 Sep 9;138(4):891-899. doi: 10.3171/2022.7.JNS22813. Print 2023 Apr 1. PMID 36087316
- [Derived] Magro E, Gentric JC, Batista AL, Kotowski M, Chaalala C, Roberge D, Weill A, Stapf C, Roy D, Bojanowski MW, Darsaut TE, Klink R, Raymond J. The Treatment of Brain AVMs Study (TOBAS): an all-inclusive framework to integrate clinical care and research. J Neurosurg. 2018 Jun;128(6):1823-1829. doi: 10.3171/2017.2.JNS162751. Epub 2017 Sep 1. PMID 28862547
- [Derived] Magro E, Gentric JC, Darsaut TE, Batista AL, Chaalala C, Roberge D, Weill A, Roy D, Bojanowski MW, Raymond J. [Treatment of brain AVMS (TOBAS): A randomized controlled trial and registry]. Neurochirurgie. 2016 Aug;62(4):197-202. doi: 10.1016/j.neuchi.2015.12.008. Epub 2016 May 25. French. PMID 27236732
- [Derived] Darsaut TE, Magro E, Gentric JC, Batista AL, Chaalala C, Roberge D, Bojanowski MW, Weill A, Roy D, Raymond J. Treatment of Brain AVMs (TOBAS): study protocol for a pragmatic randomized controlled trial. Trials. 2015 Nov 4;16:497. doi: 10.1186/s13063-015-1019-0. PMID 26530856